CLINICAL TRIAL: NCT03082170
Title: Quality of Postoperative Swallowing After Tongue Base and Palate Surgeries for Obstructive Sleep Apnea.
Brief Title: The Effect of Obstructive Sleep Apnea Operations on the Swallowing Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0587-16-RMB
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Dysphagia; Sleep Apnea, Obstructive
Keywords: sleep apnea; robotic surgery for base of tongue; soft palate surgery; post operative swallowing evaluation; dysphagia
MeSH Terms: conditions — Deglutition Disorders; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: The investigators would appreciate the quality of swallowing of participants suffering from sleep apnea that had half a year ago or more robotic resection of tongue base or soft palate surgery. The investigators will use the SDQ self reported questionnaire and the FEES test as tools for assessing the participant's swallowing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Data review (Other): The investigators will go over the data from the test summary of participants who have already undergone post operative swallowing assessment.
  Interventions: Behavioral: data review
- FEES and SDQ (Experimental): The participants will undergo six months or more after surgery swallowing assessment which will include the FEES test and the SDQ questionnaire.
  Interventions: Device: FEES; Diagnostic Test: SDQ

INTERVENTIONS:
Device: FEES — FEES test. During this test the investigators look at the pharynx and larynx of the participant while he eats and drinks Economy using number of textures aim to identify swallowing pathology.
  Arms: FEES and SDQ
Diagnostic Test: SDQ — The participant will fill a questionnaire containing 14 questions.These Questions rigorously test all aspects of the swallowing. High score in this test is consistent with swallowing disorder.
  Arms: FEES and SDQ
Behavioral: data review — Reviewing the data from the test summary of participants who have already undergone post operative swallowing assessment.
  Arms: Data review

SUMMARY:
The investigators hypothesize that partial robotic tongue base resection surgery and / or soft palate surgery, as a treatment for sleep apnea affect the swallowing quality.In order to characterize the dysphagia The investigators will locate participants undergoing this surgery more than six months ago.The investigators will test their swallowing by fiberoptic endoscopic evaluation of swallowing (FEES) and let participants fill out a questionnaire regarding swallowing disorders swallowing dysfunction questionnaire (SDQ). Also the investigators will use data collected from participants who have undergone this surgery and already had these tests due to swallowing complaints.

DETAILED DESCRIPTION:
first step: The investigators will review the operating room reports, identify participants who underwent trans-oral robotic surgery for base of tongue and/ or soft palate surgery more than six months ago.

second step:

1. The investigators will locate and conclude data of participants who already underwent assessment of postoperative swallowing function (FEES test and SDQ).The investigators will review the summary of their meeting.
2. The investigators will Call participants who have not yet done swallowing assessment and invite them to a clinic appointment.

third step- participants come to the clinic. Receive an explanation, sign a consent form. Then the participants fulfill the SDQ questionnaire (patient self- filling questionnaire) in which the participants assess the quality swallowing.

Then the investigators will conduct the swallowing test - FEES test. During This test fiber optic fiber is inserted through the participants nose for the purpose of observing the pharyngeal and laryngeal areas.The participants eat and drink food and with different textures while looking for their swallowing mechanism via the optical fiber in order to identify swallowing problems.

forth step- Two laryngologists and a speech therapists will go over the recorded swallowing tests, filling out the two questionnaires:Swallowing performance status scale (SPSS) and Penetration- aspiration scale (PAS).

With these scales every participant receives a score that reflects the quality of swallowing. A higher score indicates a more severe swallowing disorder.

ELIGIBILITY:
Inclusion Criteria:

* participants above 18 years who had Robotic base of tongue surgery and/or soft palate surgery as a treatment for obstructive sleep apnea.

Exclusion Criteria:

* participants who previously underwent surgery or treatments known to be hazardous for swallowing.
* participants suffering from a neurological problem that affects the quality of swallowing.
* Tracheostomized participants.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2017-11-20 (Estimated); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
SDQ | Six months post op
  Examination of test scores received in the SDQ
penetration aspiration scale | Six months post operative
  Examination of test scores received in the penetration aspiration scale
swallowing performance status scale | Six months post operative
  Examination of test scores received in the swallowing performance status scale

CONTACTS AND LOCATIONS:
Overall Officials: Norberto krivoy, MD, Study Chair — Rambam medical center. Haifa Israel

IPD SHARING:
Plan to Share IPD: Undecided
The data collected are summarized information regarding the swallowing quality of patients as recorded in the FEES test and as reported by the patient in the SDQ questionnaire.